CLINICAL TRIAL: NCT03844295
Title: Upper AIRway Implanted Nerve STIMulation Therapy: A Breakthrough in Obstructive Sleep Apnea Therapy
Brief Title: Obstructive Sleep Apnea Therapy by Stimulation of the Hypoglossal Nerve
Acronym: AIRSTIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Inspire Medical Systems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 38RC18.030
Record Dates: First submitted 2018-10-18; First posted 2019-02-18 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Obstructive Sleep Apnea Syndrome
Keywords: stimulation; hypoglossal nerve; Upper-airway
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: Monocentric, prospective, controlled, patient single-blind study
Who Masked: Participant
Masking Description: Only patient will be blind. He doesn't know if INSPIRE therapy was activated or not
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Activated Inspire® Upper Airway Stimulation System (Experimental): INSPIRE® device will be active a month
  Interventions: Device: Activated Inspire® Upper Airway Stimulation System
- Inactivated Inspire® Upper Airway Stimulation System (Placebo Comparator): After a period 15 days of "wash-out" the INSPIRE® device will be inactivated for a second period of one month.
  Interventions: Device: Inactivated Inspire® Upper Airway Stimulation System

INTERVENTIONS:
Device: Activated Inspire® Upper Airway Stimulation System — At first, INSPIRE® device will be active a month
  Arms: Activated Inspire® Upper Airway Stimulation System
Device: Inactivated Inspire® Upper Airway Stimulation System — After 15 days "wash-out" INSPIRE® device will be inactivated for a second period of one month.
  Arms: Inactivated Inspire® Upper Airway Stimulation System

SUMMARY:
Continuous positive airway pressure (CPAP) is the gold standard to normalize breathing during sleep in patients with obstructive sleep apnea syndrom (OSA). Many patients will not tolerate or will not accept CPAP. Implanted nerve stimulation is a novel therapy for OSA patients that restores the upper airway potency using unilateral XII nerve electric stimulation.

The principal objective of this study is short-term efficacy of a new treatment for OSA on blood pressure variability during sleep.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) syndrome had become over the last decade a serious health concern due to its high prevalence which raise 10% of the general population.

It is characterized by recurrent episodes of airflow obstruction in the upper airway (UA) consequence of passive collapse of the UA, particularly at the tongue level. These collapses induce recurrent asphyxia that results in oxygen desaturations with persistant and crescendo respiratory efforts inducing arousals from sleep.

Indeed, despite its large efficacy some of the patients will never accept continuous positive airway pressure treatment or will not tolerate. To this extent, alternative treatement has been developed: implanted hypoglossal stimulation. This treatment has been developed by Inspire Medical Device. The Inspire® system is intended to prevent base-of-tongue obstruction as well as specific soft palate obstructions by stimulating the hypoglossal nerve synchronous with respiration.

A selection processus will be applied in order to identify the patients that will be good responders to the hypoglossal stimulation.

The main criterion of selection is based on Drug Induced Sleep Endoscopy(DISE) that will be performed by a trained endoscopist dedicated to this study.

This sleep endoscopy allows to visualize during induced sleep the shape of the UA and the type of collapsus. Indeed an antero-posterior collapsus is related to a good response to hypoglossal nerve stimulation while complete concentric obstruction at velopharyngeal is a predictor of poor response.

In this pilot study, the investigators evaluate as a primary outcome the delta range of blood pressure during sleep but also other cardiovascular indexes targeting blood pressure and heart rate variability as secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 to 80 years old
* Patient with moderate to severe OSA based on an established diagnosis of OSA (15≤AHI<65) by polysomnography or respiratory polygraphy not older thant three years.
* Patient with moderate to severe OSA naïve of treatment or with difficulty accepting or adhering to CPAP treatment.
* Willing and capable to have stimulation hardware permanently implanted, and to use the patient programmer to activate the stimulation
* Willing and capable to return for all follow-up visits and conduct sleep studies at home, including the evaluation procedures and filling out questionnaires
* Willing and capable of providing written informed consent.

Exclusion Criteria:

* Any anatomical finding that would compromise the performance of upper airway stimulation, such as the presence of complete concentric collapse of the soft palate
* Have any condition or procedure that has compromised neurological control of the upper airway
* Unable to operate the patient programmer
* Pregnant or plan to become pregnant, and breastfeeding women
* Require magnetic resonance imaging (MRI)
* Have an implantable device that may be susceptible to unintended interaction with the Inspire system.

Additional exclusions for study purposes only

* Body Mass Index (BMI) of >32
* Central + mixed apneas > 25% of the total apnea-hypopnea index (AHI)
* Neuromuscular disease
* Hypoglossal-nerve palsy
* Severe restrictive or obstructive pulmonary disease
* Moderate-to-severe pulmonary arterial hypertension
* Severe valvular heart disease
* New York Heart Association class III or IV heart failure
* Recent myocardial infarction or severe cardiac arrhythmias (within the past 6 months)
* Persistent uncontrolled hypertension despite medication use
* Coexisting nonrespiratory sleep disorders that would confound functional sleep assessment
* Any chronic medical illness or condition that contraindicates a surgical procedure under general anesthesia, as judged by the clinical study Investigator
* a terminal illness with life expectancy < 12 months
* Active psychiatric disease (psychotic illness, major depression, or acute anxiety attacks) which prevents subject compliance with the requirements of the investigational study testing
* Radiotherapy or ablation therapy of the head and/or neck
* Surgical resection for cancer or congenital malformations in the larynx, tongue, or throat(with exception of tonsillectomy and/or adenoidectomy)
* Previous surgery within 3 months performed on the soft-palate tissue
* Obvious fixed upper airway obstructions (tumors, polyps, unilateral nasal obstruction)
* Need for chronic supplemental oxygen therapy for any other reason, pO2 (partial pressure of oxygen) < 55 mm Hg
* Clinical evidence of severe renal failure (Stage 4 or 5) undergoing dialysis or expected to institute dialysis within 6 months
* Patients on medication that may alter consciousness, the pattern of respiration or sleep architecture (for example, benzodiazepiones, opiates, neuroleptics, prescription stimulants, phenothiazine, or any form of chemical substance abuse)
* Patients taking blood thinning medications (for example warfarin, aspirin, plavix or other blood thinning agents which cannot be safety stopped or bridged temporarily to allow surgery to take place)
* Any other reason for the investigator deems that the subject is unfit for participation in the study
* Subject in exclusion period for another study
* Subject under administrative or judicial control.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-03-21 (Actual); Primary Completion 2021-12-22 (Actual); Study Completion 2023-10-10 (Actual)

PRIMARY OUTCOMES:
Short-term efficacy of a new treatment for OSA on systolic blood pressure variability during sleep | one month treatment active versus non active treatment
  Change in the difference between delta nocturnal systolic blood pressure (difference between maximum and minimal nocturnal systolic blood pressure ; nocturnal period is defined from 10 pm to 7am).

SECONDARY OUTCOMES:
Short-term efficacy of a new treatment for OSA on mean-24h, daytime and nighttime blood pressure | one month treatment active versus non active treatment
  Ambulatory 24h arterial blood pressure
Clinical efficacy of this new treatment on OSA by Epworth sleepiness scale score | one month treatment active versus non active treatment
  It's a self-administered questionnaire with 8 questions. Patients are asked to rate, on a 4-point scale (0-3), their usual chances of dozing off or falling asleep while engaged in eight different activities. The ESS score (the sum of 8 item scores, 0-3) can range from 0 to 24. The higher the ESS score, the higher that person has daytime sleepiness.
Clinical efficacy of this new treatment on Apnea-Hypopnea Index measured by polysomnography | one month treatment active versus non active treatment
  Apnea-Hypopnea Index expressed in number per hour
Change in sympatho-vagal balance based on heart rate variability analysis | one month treatment active versus non active treatment
  ECG polysomnography
Self-reported changes in sleep and quality of life by SF-36 score | one month treatment active versus non active treatment
  The SF-36 is a 36-item scale constructed to survey health status and quality of life (Ware & Sherbourne, 1992), assessing eight health concepts: limitations in Quality of life physical activities because of health problems; limitations in social activities because of physical or emotional problems; limitations in usual role activities because of physical health problems); bodily pain; general mental health (psychological distress and well-being); limitations in usual role activities because of emotional problems; vitality (energy and fatigue); and general health perceptions. The standard form of the instruments asks for participants to reply to questions according to how they have felt over the previous week. The items use Likert-type scales, some with 5 or 6 points and others with 2 or 3 points. The SF-36 has been widely used and has excellent psychometrics.
Sleep latency assessed during a Maintenance of Wakefulness Test | one month treatment active versus non active treatment
  Mean sleep latency from the 4 sessions of the Maintenance of Wakefulness Test
Nocturnal pulse pressure assessed by Continuous Non-invasive Arterial Pressure monitoring | one month treatment active versus non active treatment
  Pulse pressure variability indexe DeltaBP in mmHg.
Short-term efficacy of a new treatment for OSA on diastolic blood pressure variability during sleep | one month treatment active versus non active treatment
  Change in the difference between delta nocturnal systolic blood pressure (difference between maximum and minimal nocturnal systolic blood pressure ; nocturnal period is defined from 10 pm to 7am).
Clinical efficacy of this new treatment on OSA by Pichot weakness scale score | one month treatment active versus non active treatment
  It's a self-administered questionnaire with 8 questions. Patients are asked to rate, on a 5-point scale (0-4), their usual feeling of tiredness or weakness while engaged in eight different activities. The PWS score (the sum of 8 item scores, 0-4) can range from 0 to 32. The higher the PWS score, the higher that person has weakness.
Clinical efficacy of this new treatment on nocturia | one month treatment active versus non active treatment
  Assessment of nocturia number by nigt
Clinical efficacy of this new treatment on morning asthenia | one month treatment active versus non active treatment
  Patients are asked to assess, on a visual analogic scale morning asthenia. The items use a visual analogic scales from 0 to 10 points.
Clinical efficacy of this new treatment on morning headache | one month treatment active versus non active treatment
  Patients are asked to assess, on a visual analogic scale morning headache. The items use a visual analogic scales from 0 to 10 points.
Clinical efficacy of this new treatment on snoring | one month treatment active versus non active treatment
  Patients are asked to assess, on a visual analogic scale snoring. The items use a visual analogic scales from 0 to 10 points.
Self-reported changes in sleep and quality of life by FOSQ score | one month treatment active versus non active treatment
  This is a disease specific quality of life questionnaire to determine functional status in adults; measures are designed to assess the impact of disorders of excessive sleepiness on multiple activities of everyday living and the extent to which these abilities are improved by effective treatment. The 5 domains that the FOSQ measures are as follows: Activity level, vigilance, intimacy and sexual relationships, general productivity, social outcome, rate the difficulty of performing a given activity on a 4-point scale (no difficulty to extreme difficulty).
Clinical efficacy of this new treatment on oxygen desaturation index measured by polysomnography | one month treatment active versus non active treatment
  Oxygen desaturation index expressed in number
Clinical efficacy of this new treatment on sleep efficacy measured by polysomnography | one month treatment active versus non active treatment
  Sleep efficacy expressed by ratio of total sleep time on total sleep period

CONTACTS AND LOCATIONS:
Overall Officials: Renaud RT TAMISIER, PhD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- UniversityHospitalGrenoble, Grenoble, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Young T, Palta M, Dempsey J, Skatrud J, Weber S, Badr S. The occurrence of sleep-disordered breathing among middle-aged adults. N Engl J Med. 1993 Apr 29;328(17):1230-5. doi: 10.1056/NEJM199304293281704. PMID 8464434
- [Background] Young T, Peppard PE, Gottlieb DJ. Epidemiology of obstructive sleep apnea: a population health perspective. Am J Respir Crit Care Med. 2002 May 1;165(9):1217-39. doi: 10.1164/rccm.2109080. PMID 11991871
- [Background] Mulgrew AT, Ryan CF, Fleetham JA, Cheema R, Fox N, Koehoorn M, Fitzgerald JM, Marra C, Ayas NT. The impact of obstructive sleep apnea and daytime sleepiness on work limitation. Sleep Med. 2007 Dec;9(1):42-53. doi: 10.1016/j.sleep.2007.01.009. Epub 2007 Sep 6. PMID 17825611
- [Background] Lallukka T, Kaikkonen R, Harkanen T, Kronholm E, Partonen T, Rahkonen O, Koskinen S. Sleep and sickness absence: a nationally representative register-based follow-up study. Sleep. 2014 Sep 1;37(9):1413-25. doi: 10.5665/sleep.3986. PMID 25142569
- [Background] Tamisier R, Pepin JL, Remy J, Baguet JP, Taylor JA, Weiss JW, Levy P. 14 nights of intermittent hypoxia elevate daytime blood pressure and sympathetic activity in healthy humans. Eur Respir J. 2011 Jan;37(1):119-28. doi: 10.1183/09031936.00204209. Epub 2010 Jun 4. PMID 20525723
- [Background] Pepin JL, Tamisier R, Barone-Rochette G, Launois SH, Levy P, Baguet JP. Comparison of continuous positive airway pressure and valsartan in hypertensive patients with sleep apnea. Am J Respir Crit Care Med. 2010 Oct 1;182(7):954-60. doi: 10.1164/rccm.200912-1803OC. Epub 2010 Jun 3. PMID 20522795
- [Background] Gagnadoux F, Fleury B, Vielle B, Petelle B, Meslier N, N'Guyen XL, Trzepizur W, Racineux JL. Titrated mandibular advancement versus positive airway pressure for sleep apnoea. Eur Respir J. 2009 Oct;34(4):914-20. doi: 10.1183/09031936.00148208. Epub 2009 Mar 26. PMID 19324954
- [Background] Strollo PJ Jr, Soose RJ, Maurer JT, de Vries N, Cornelius J, Froymovich O, Hanson RD, Padhya TA, Steward DL, Gillespie MB, Woodson BT, Van de Heyning PH, Goetting MG, Vanderveken OM, Feldman N, Knaack L, Strohl KP; STAR Trial Group. Upper-airway stimulation for obstructive sleep apnea. N Engl J Med. 2014 Jan 9;370(2):139-49. doi: 10.1056/NEJMoa1308659. PMID 24401051
- [Background] Mayer P, Pepin JL, Bettega G, Veale D, Ferretti G, Deschaux C, Levy P. Relationship between body mass index, age and upper airway measurements in snorers and sleep apnoea patients. Eur Respir J. 1996 Sep;9(9):1801-9. doi: 10.1183/09031936.96.09091801. PMID 8880094
- [Background] Eastwood PR, Barnes M, Walsh JH, Maddison KJ, Hee G, Schwartz AR, Smith PL, Malhotra A, McEvoy RD, Wheatley JR, O'Donoghue FJ, Rochford PD, Churchward T, Campbell MC, Palme CE, Robinson S, Goding GS, Eckert DJ, Jordan AS, Catcheside PG, Tyler L, Antic NA, Worsnop CJ, Kezirian EJ, Hillman DR. Treating obstructive sleep apnea with hypoglossal nerve stimulation. Sleep. 2011 Nov 1;34(11):1479-86. doi: 10.5665/sleep.1380. PMID 22043118
- [Background] Goding GS Jr, Tesfayesus W, Kezirian EJ. Hypoglossal nerve stimulation and airway changes under fluoroscopy. Otolaryngol Head Neck Surg. 2012 Jun;146(6):1017-22. doi: 10.1177/0194599812436472. Epub 2012 Feb 3. PMID 22307575
- [Background] Schwartz AR, Barnes M, Hillman D, Malhotra A, Kezirian E, Smith PL, Hoegh T, Parrish D, Eastwood PR. Acute upper airway responses to hypoglossal nerve stimulation during sleep in obstructive sleep apnea. Am J Respir Crit Care Med. 2012 Feb 15;185(4):420-6. doi: 10.1164/rccm.201109-1614OC. Epub 2011 Dec 1. PMID 22135343
- [Background] Mwenge GB, Dury M, Delguste P, Rodenstein D. Response of automatic continuous positive airway pressure devices in a normal subject. Eur Respir J. 2011 Jun;37(6):1530-3. doi: 10.1183/09031936.00139510. No abstract available. PMID 21632834
- [Background] Oldenburg O, Lamp B, Faber L, Teschler H, Horstkotte D, Topfer V. Sleep-disordered breathing in patients with symptomatic heart failure: a contemporary study of prevalence in and characteristics of 700 patients. Eur J Heart Fail. 2007 Mar;9(3):251-7. doi: 10.1016/j.ejheart.2006.08.003. Epub 2006 Oct 5. PMID 17027333
- [Background] Somers VK, Dyken ME, Clary MP, Abboud FM. Sympathetic neural mechanisms in obstructive sleep apnea. J Clin Invest. 1995 Oct;96(4):1897-904. doi: 10.1172/JCI118235. PMID 7560081
- [Background] Tamisier R, Tan CO, Pepin JL, Levy P, Taylor JA. Blood Pressure Increases in OSA due to Maintained Neurovascular Sympathetic Transduction: Impact of CPAP. Sleep. 2015 Dec 1;38(12):1973-80. doi: 10.5665/sleep.5252. PMID 26039959
- [Background] Berry RB, Budhiraja R, Gottlieb DJ, Gozal D, Iber C, Kapur VK, Marcus CL, Mehra R, Parthasarathy S, Quan SF, Redline S, Strohl KP, Davidson Ward SL, Tangredi MM; American Academy of Sleep Medicine. Rules for scoring respiratory events in sleep: update of the 2007 AASM Manual for the Scoring of Sleep and Associated Events. Deliberations of the Sleep Apnea Definitions Task Force of the American Academy of Sleep Medicine. J Clin Sleep Med. 2012 Oct 15;8(5):597-619. doi: 10.5664/jcsm.2172. PMID 23066376